CLINICAL TRIAL: NCT02114645
Title: To Evaluate the Effect of GnRH Agonist Administered in the Luteal Phase on ART Cycle Outcomes in Both GnRH Agonist and GnRH Antagonist Treated Ovarian Stimulation Protocols
Brief Title: The Effect of GnRH Agonist Administered in the Luteal Phase on ART Cycle Outcomes
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Zekai Tahir Burak Women's Health Research and Education Hospital (Other)
Responsible Party: Principal Investigator, Nagihan CENGAVER, Resident, Zekai Tahir Burak Women's Health Research and Education Hospital
Allocation: Non-Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: ZTB-5030; ZTB5030 (Registry Identifier: ZekaiTahirBurak)
Record Dates: First submitted 2014-04-08; First posted 2014-04-15 (Estimated); Last update posted 2014-04-15 (Estimated); Status verified 2014-04

CONDITIONS: Infertility
Keywords: Luteal phase support,GnRH agonist,ART cycles
MeSH Terms: conditions — Infertility | interventions — Leuprolide; Estradiol; estradiol, estriol drug combination; Tablets

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- LongGnRH agonist protocol(controlgroup) (Active Comparator): Long GnRH agonist protocol ( control group) Luteal Phase Support: Vaginal progesterone + 4mg oral estradiol valerate
  Interventions: Drug: vaginal progesterone; Drug: 4 mg oral estradiol valerate
- Long protocol-leuprolide acetate (Experimental): Long GnRH agonist protocol Luteal Phase Support: Vaginal progesterone+oral estradiol valerate subcutaneous 0.5mg leuprolide acetate fifth and tenth day after embryo transfer
  Interventions: Drug: Leuprolide acetate; Drug: vaginal progesterone; Drug: 4 mg oral estradiol valerate
- GnRHantagonist protocol(control group) (Active Comparator): GnRH antagonist protocol ( control group) Luteal Phase Support: Vaginal progesterone + 4mg oral estradiol valerate
  Interventions: Drug: vaginal progesterone; Drug: 4 mg oral estradiol valerate
- antagonist protocol-leuprolide acetate (Experimental): GnRH antagonist protocol Luteal Phase Support: Vaginal progesterone + 4mg oral estradiol valerate + subcutaneous 0.5mg leuprolide acetate fifth and tenth day after embryo transfer
  Interventions: Drug: Leuprolide acetate; Drug: vaginal progesterone; Drug: 4 mg oral estradiol valerate

INTERVENTIONS:
Drug: Leuprolide acetate — in experimentals groups,on fifth and tenth day after embryo transfer 0,5mg leuprolide acetate is given subcutaneously as luteal phase support
  Other Names: lucrin
  Arms: Long protocol-leuprolide acetate; antagonist protocol-leuprolide acetate
Drug: vaginal progesterone — crinone gel is applied till fetal heart beat is detected
  Other Names: crinone gel
Drug: 4 mg oral estradiol valerate — estrofem is given twice a day
  Other Names: estrofem 2mg tablet

SUMMARY:
This prospective clinical trial evaluates the effect of a two dose GnRH agonist administered in the luteal phase on the outcome of ART cycles stimulated with the long GnRH agonist and GnRH antagonist protocol.

DETAILED DESCRIPTION:
This prospective clinical trial evaluates the effect of a two dose GnRH agonist administered in the luteal phase on the outcome of ART cycles stimulated with the long GnRH agonist and GnRH antagonist protocol. Decision between each of these two protocols was subjective and depended on the clinical context.In addition to routine luteal phase support with progesterone and estradiol valerate,women received two dose of GnRH agonist on the fifth and tenth day after ET.Live birth rate was the primary outcome measure.

ELIGIBILITY:
Inclusion Criteria:

* Couples undergoing ART with their own gametes.
* Couples having at least one good embryo available for transfer.
* Normoresponder
* Infertility etiology is unexplained
* ovulation triggered by intramuscular injection of 10000 IU of HCG

Exclusion Criteria:

Patients older than 38 years old

* High and poor responder patients

Ages: 18 Years to 38 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 2014-04; Primary Completion 2015-02 (Estimated); Study Completion 2015-04 (Estimated)

PRIMARY OUTCOMES:
Live Birth Rate | 42 weeks

SECONDARY OUTCOMES:
Ongoing pregnancy | more than 20 weeks
miscarriage | up to 20 weeks
OHSS | up to 10 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Nagihan Cengaver, Resident, Principal Investigator — Zekai Tahir Burak Women's Health Research and Education Hospital
Locations (1):
- Zekai Tahir Burak Hospital, Ankara, Cankaya, Turkey (Türkiye)

REFERENCES:
- See also: Beneficial effect of luteal-phase GnRH agonist administration on embryo implantation after ICSI in both GnRH agonist- and antagonist-treated ovarian stimulation cycles. — http://www.ncbi.nlm.nih.gov/pubmed/?term=16926261